CLINICAL TRIAL: NCT02604004
Title: Bioequivalence Study Between Lamivudine Formulations in the Form of Coated Tablet 150 mg (Test) and EPIVIR of Glaxosmithkline in Healthy Volunteers of Both Genders in Fasting Condition
Brief Title: Bioequivalence Study Between Lamivudine Formulations in the Form of Coated Tablet of 150 mg in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, José Homero de Souza Filho, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NUD_04_12
Record Dates: First submitted 2015-11-05; First posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: HIV INFECTIONS
Keywords: lamivudine; bioequivalence test; pharmacokinetics; high-performance liquid chromatography; 3TC; LC-MS/MS; mass spectrometry
MeSH Terms: conditions — HIV Infections | interventions — Lamivudine; Tablets; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Period 1 (Active Comparator): Epivir ® tablet 150-mg single dose (drug reference)
  Interventions: Drug: Epivir ® tablet 150-mg single dose (drug reference); Drug: Lamivudine 150-mg tablet single dose (drug test)
- Period 2 (Experimental): Lamivudine 150-mg tablet single dose (drug test)
  Interventions: Drug: Epivir ® tablet 150-mg single dose (drug reference); Drug: Lamivudine 150-mg tablet single dose (drug test)

INTERVENTIONS:
Drug: Epivir ® tablet 150-mg single dose (drug reference) — Bioequivalence lamivudine 150 mg tablets fasting condition
  Other Names: lamivudine; 3TC
Drug: Lamivudine 150-mg tablet single dose (drug test) — Bioequivalence lamivudine 150 mg tablets fasting condition
  Other Names: 3TC

SUMMARY:
The objective of this research is to check whether the test drug (lamivudine in the form of coated tablet 150 mg) achieves plasma levels equivalent to those obtained from the EPIVIR in the form of coated tablet 150 mg GlaxoSmithKline administered to 28 volunteers of both genres under fasting condition.

DETAILED DESCRIPTION:
It is an open, randomized, crossover 2x2, single dose, with the administration of medicine with 28 healthy volunteers, adults aged 18-50 years, of both genders (14 males and 14 females). Of the 28 volunteers planned in the study protocol to start, gave up one (woman) before the start of Phase I. So the study was initiated and completed with the participation of 27 volunteers. The volunteers were in hospital for a period of approximately 36 hours in each stage.

ELIGIBILITY:
Inclusion Criteria:

* Considered healthy after undergoing a clinical evaluation;
* Agree freely and sign the Recruitment and Informed Consent Term, after all the content of the protocol was clear before any procedure;
* Present the body mass index greater than 19 and less than 30.

Exclusion Criteria:

* Results of laboratory tests outside the range considered normal, unless they were considered clinically irrelevant;
* Allergic to lamivudine or any other drug;
* Positive outcome of the pre-admission pregnancy test;
* Regular medication within four (4) weeks prior to the start of the study or use of any medication to present interaction with lamivudine one week before the start of the study;
* Use abusive alcoholic beverage;
* Use of illicit drugs and tobacco;
* History of liver disease, renal, pulmonary, gastrointestinal, epileptic, hematologic or psychiatric; hypo- or hypertension of any cause that required pharmacological treatment; myocardial infarction, angina and / or heart failure;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
AUClast | Up to 36 hours
  Area under the Plasma concentration-time curve from time Zero to last time (AUCinf) of lamivudine in plasma.

SECONDARY OUTCOMES:
Cmax | Up to 36 hours
  Maximum concentration (Cmax) of lamivudine in plasma.
Tmax | Up to 36 hours
  Time for Maximum concentration (Tmax) of lamivudine in plasma.
T1/2 | Up to 72 hours
  Terminal half-time of lamivudine in plasma.
AUCinf | Up to 36 hours
  Area under the Plasma concentration-time curve from time Zero to infinity (AUCinf) of lamivudine in plasma.

REFERENCES:
- [Result] Goodman & Gilman's The Pharmacologic Basis of Therapeutics - 11th Ed. (2006)
- [Result] Martindale The Complete Drug Reference - Thirty-sixth edition (2009).
- [Result] http://www4.anvisa.gov.br/base/visadoc/BM/BM[25676-1-0].PDF acessado em 13/10/2011.
- [Result] ANVISA. Manual de Boas Práticas em Biodisponibilidade/ Bioequivalência. Volume I. Agência Nacional de Vigilância Sanitária. Brasília: ANVISA, 2002.
- [Result] ANVISA. Resolução RE nº 899, de 29 de maio de 2003. "Guia para validação de métodos analíticos e bioanalíticos". ANVISA-MS, Brasília.
- [Result] ANVISA. Resolução RE nº 1170, de 19 de abril de 2006. "Guia para provas de biodisponibilidade relativa/ bioequivalência de medicamentos". ANVISA-MS, Brasília.
- [Result] ANVISA. "Guia para planejamento e realização da etapa estatística de estudos de Biodisponibilidade relativa / Bioequivalência". RE Nº. 898, de 29 de maio de 2003.
- [Result] Kano EK, dos Reis Serra CH, Koono EE, Andrade SS, Porta V. Determination of lamivudine in human plasma by HPLC and its use in bioequivalence studies. Int J Pharm. 2005 Jun 13;297(1-2):73-9. doi: 10.1016/j.ijpharm.2005.03.002. Epub 2005 Apr 26. PMID 15907596
- [Result] Narang VS, Lulla A, Malhotra G, Purandare S. Pharmacokinetic profiling and bioequivalence evaluation of 2 lamivudine tablet formulations after single oral administration in healthy human Indian volunteers. J Acquir Immune Defic Syndr. 2005 Apr 15;38(5):566-9. doi: 10.1097/01.qai.0000155202.51232.f5. PMID 15793367
- [Result] Schwartz JB. The influence of sex on pharmacokinetics. Clin Pharmacokinet. 2003;42(2):107-21. doi: 10.2165/00003088-200342020-00001. PMID 12537512
- [Result] Wald A, Van Thiel DH, Hoechstetter L, Gavaler JS, Egler KM, Verm R, Scott L, Lester R. Gastrointestinal transit: the effect of the menstrual cycle. Gastroenterology. 1981 Jun;80(6):1497-500. PMID 7227774
- [Result] Greenblatt DJ, Divoll M, Harmatz JS, Shader RI. Oxazepam kinetics: effects of age and sex. J Pharmacol Exp Ther. 1980 Oct;215(1):86-91. PMID 7452494
- [Result] FLOCKHART D. A. Drug interactions: Cytochrome P450 drug interaction table. Indiana School of Medicine. 2007. http://medicine.iupui.edu/clinpharm/ddis/ table.asp. Accessed December 1, 2009.
- [Result] Bigos KL, Pollock BG, Stankevich BA, Bies RR. Sex differences in the pharmacokinetics and pharmacodynamics of antidepressants: an updated review. Gend Med. 2009 Dec;6(4):522-43. doi: 10.1016/j.genm.2009.12.004. PMID 20114004
- [Result] Ofotokun I, Chuck SK, Hitti JE. Antiretroviral pharmacokinetic profile: a review of sex differences. Gend Med. 2007 Jun;4(2):106-19. doi: 10.1016/s1550-8579(07)80025-8. PMID 17707845
- [Result] Pluda JM, Cooley TP, Montaner JS, Shay LE, Reinhalter NE, Warthan SN, Ruedy J, Hirst HM, Vicary CA, Quinn JB, et al. A phase I/II study of 2'-deoxy-3'-thiacytidine (lamivudine) in patients with advanced human immunodeficiency virus infection. J Infect Dis. 1995 Jun;171(6):1438-47. doi: 10.1093/infdis/171.6.1438. PMID 7769277
- [Result] van Leeuwen R, Katlama C, Kitchen V, Boucher CA, Tubiana R, McBride M, Ingrand D, Weber J, Hill A, McDade H, et al. Evaluation of safety and efficacy of 3TC (lamivudine) in patients with asymptomatic or mildly symptomatic human immunodeficiency virus infection: a phase I/II study. J Infect Dis. 1995 May;171(5):1166-71. doi: 10.1093/infdis/171.5.1166. PMID 7751691
- [Result] Johnson MA, Moore KH, Yuen GJ, Bye A, Pakes GE. Clinical pharmacokinetics of lamivudine. Clin Pharmacokinet. 1999 Jan;36(1):41-66. doi: 10.2165/00003088-199936010-00004. PMID 9989342
- [Result] Perry CM, Faulds D. Lamivudine. A review of its antiviral activity, pharmacokinetic properties and therapeutic efficacy in the management of HIV infection. Drugs. 1997 Apr;53(4):657-80. doi: 10.2165/00003495-199753040-00008. PMID 9098665
- [Result] World Medical Association Declaration of Helsinki (WMA). Ethical Principles for Medical Research Involving Human Subjects. Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the 52nd WMA General Assembly, Edinburgh, Scotland, October 7, 2000 [WMA Web site]. http://www.wma.net/e/policy/b3.htm . Accessed December 20, 2009
- [Result] Center for Drug Evaluation and Research, US Food and Drug Administration. Guidance for Industry: Bioavailability and Bioequivalence Studies for Orally Administered Drug Products-General Considerations [COER Web site). http://www.fda.gov/cder/guidance/5356ful.pdf. Accessed February 22, 2010.
- [Result] EMEA (European Agency for the Evaluation of Medicinal Products). CPMP (Committee for Propietary Medicinal Products). Note for guidance on the investigation of bioavailability and bioequivalence. London, July 2001.